CLINICAL TRIAL: NCT03307668
Title: Study on Efficacy and Safety of CaReSR-1S to Repair Cartilage Defects of the Knee: a Randomised, Multicentre, Open-label, Controlled Trial
Brief Title: Study on Efficacy and Safety of CaReSR-1S to Repair Cartilage Defects of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arthro-Anda Tianjin Biologic Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.0
Record Dates: First submitted 2017-08-24; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Cartilage Defects
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaReS-1S (Experimental)
  Interventions: Device: CaReSR-1S
- Microfracture (Active Comparator)
  Interventions: Device: Microfracture

INTERVENTIONS:
Device: CaReSR-1S — CaReSR-1S is a sterile, ready for use round implant based on a dense matrix of native Collagen type I.
  Arms: CaReS-1S
Device: Microfracture — Microfracture is an articular cartilage repair surgical technique that works by creating tiny fractures in the underlying bone. This causes new cartilage to develop from a so-called super-clot.
  Arms: Microfracture

SUMMARY:
The purpose of this trial is to investigate the safety and effect of CaReS-1S to repair knee cartilage defects.

DETAILED DESCRIPTION:
CaReSR-1S is a sterile, ready for use round implant based on a dense matrix of native Collagen type I. It is indicated for the defect filling of focal, full layer and clearly defined knee and ankle cartilage defects of longest diameter 1.1-2.2cm. The fixation of CaReSR-1S is made for all sizes with fibrin glue, whereas the 11 mm implants also allow a press-fit anchoring due to the elasticity of the implant.

The physical nature of the CaReSR-1S allows the in-growth of healthy chondrocytes, as well as progenitor cells from the surrounding healthy tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 55 years old;
2. Diagnosed with isolated knee cartilage defects in condyles of femur by arthroscopy, and the longest diameter is 1.1-2.2cm. The degree of the cartilage defects is Outerbridge IV degree or III degree but approximate to IV degree;
3. Outerbridge degree of cartilage in the other articular facet ≤Ⅱ;
4. Normal lower limb mechanical force line (varus or valgum < 5°);
5. Skeletal mature;
6. 18Kg/M2 ≤ BMI ≤ 30Kg/M2;
7. Agree to sign the informed consent form;
8. Can cooperate in a post-operative rehabilitation program.

Exclusion Criteria:

1. Superficial cartilage defects;
2. Concomitant with subchondral bone defect;
3. Varus or valgum > 5°;
4. Serious meniscus injury;
5. Fractures around the knee;
6. Cannot join in the post-operative rehabilitation program;
7. The contralateral lower-limb cannot stand weight-bearing;
8. A history of knee surgery within 6 months;
9. Secondary arthritis affecting cartilage;
10. Serious arthrocleisis;
11. Undergoing clinical trial;
12. Serious illness of the heart, lung, and other vital organs;
13. Liver function test equal to two times or greater than the upper normal limits; serum creatinine equal to two times or greater than the upper normal limit;
14. Have a contagious disease;
15. Allergic to the agents;
16. Lactating or pregnant women;
17. Serious neuropathy or mental disease;
18. Be addicted with drug or alcohol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of Magnetic resonance observation of cartilage repair tissue (MOCART) score between two groups | 12 months

SECONDARY OUTCOMES:
Difference of MOCART score change from baseline between groups | 12 months
Difference of International Knee Documentation Committee (IKDC) Subjective Knee Form score change from baseline between groups | 12 months
Difference of Lysholm score change from baseline between groups | 12 months
"Good""Moderate""Poor" rates according to Lysholm score | 12 months
Effective rate according to Lysholm score | 12 months
Total efficiency according to Lysholm score | 12 months
Incidence of treatment-related adverse events | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No